CLINICAL TRIAL: NCT06059521
Title: Randomized Controlled Study on Subjective Refraction by Software Eye Test Technology Versus Retinoscopy
Brief Title: Software Refraction With Mobilerone Versus Retinoscopy
Acronym: SRMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Airdoc Technology Co., Ltd. (Industry)
Collaborators: University of Notre Dame Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AirdocSoftwareEyeTest
Record Dates: First submitted 2023-07-24; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Myopia; Myopia, Moderate; Astigmatism
Keywords: software; refraction; subjective refraction; mobilerone; myopia; astigmatism
MeSH Terms: conditions — Myopia; Lymphoma, Follicular; Astigmatism | interventions — Retinoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Software Refraction (Experimental): Refraction is done by software with subjective refraction through a mobilerone.
  Interventions: Device: Software refraction with Eye Test Technology in a mobilerone
- Refraction by retinoscopy (Active Comparator): Refraction is done objectively by retinoscopy.
  Interventions: Device: Retinoscopy

INTERVENTIONS:
Device: Software refraction with Eye Test Technology in a mobilerone — Refraction is done by software App by a mobilerone software installed.
  Other Names: Online refraction or App refraction with Eye Test Technology
  Arms: Software Refraction
Device: Retinoscopy — Retinoscopy is an objective refraction method with retinoscope.
  Other Names: Refraction by retinoscopy
  Arms: Refraction by retinoscopy

SUMMARY:
Software refraction in the mobilerone for myopia and astigmatism is a novel medical device for myopia adults and elder children with or without astigmatism. And the investigators would like to test its accuracy and efficacy as well as safety.

DETAILED DESCRIPTION:
It's a software installed in a mobilerone with subjective guide on screen for testing myopic refractive error with or without astigmatism for adults or elder children. The investigators would like to compare its refraction results with retinoscopy.

ELIGIBILITY:
Inclusion Criteria:

* • subject with ametropia on each eye ≤-12.00D

  * subject with best corrected visual acuity ≥ 20/25, no amblyopia
  * subject with normal transparency of eyes
  * subject with a healthy fundus that does not reveal major abnormalities that may affect vision due to the fluctuate situations
  * subject able to cooperate with the screen and the operator
  * subject without heavy drug treatment that may affect vision as synthetic antimalarials, corticosteroids
  * non-diabetic subject
  * non nystagmus subject
  * non-strabismus subject
  * subject who has not had eye surgery less than 1 year old

Exclusion Criteria:

* • subject with a topography showing an anomaly (keratoconus type or other)

  * subject with hyperopia or presbyopia
  * subject with mild myopia ≥ -1.00D
  * subject who cannot speak with the operator including those staff of local optometrists or ophthalmologists

Ages: 10 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Spherical Equivalence(D) | 1-day and within 2 weeks
  Spherical is myopic equivalence with total spherical plus half the cylinder diopter.
Astigmatism Power(D) | 1-day and within 2 weeks
  Cylinder value of each total astigmatism power
Astigmatism axial | 1-day and within 2 weeks
  Cylinder axis of astigmatism
pupil distance (mm) | 1-day and within 2 weeks
  pupil distance measurement with software or autorefractor

SECONDARY OUTCOMES:
Efficacy of test time (minutes) | 1-day and within 2 eeks
  How long for each test

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Airdoc MPC Opthalmology Clinics, Beijing, Beijing Municipality
  - Jenny QIU, Beijing, Beijing Municipality
  - Qiu Jenny, Beijing, Haidian District

IPD SHARING:
Plan to Share IPD: No